CLINICAL TRIAL: NCT01054261
Title: A Phase I, Open-Label, Parallel-Group, Single Dose, Non-Randomized Study to Compare the Pharmacokinetics of Avanafil in Male Subjects With Mild and Moderate Renal Impairment to Subjects With Normal Renal Function
Brief Title: To Compare the Pharmacokinetics of Avanafil in Subjects With Mild and Moderate Renal Impairment to Subjects With Normal Renal Function.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wesley Day, VP Clinical Operations
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA-013
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Renal
Keywords: avanafil, renal, impairment, TA-1790
MeSH Terms: interventions — avanafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal (Other): Normal renal function
  Interventions: Drug: avanafil
- Mild (Other): Mild renal impairment
  Interventions: Drug: avanafil
- Moderate (Other): Moderate renal impairment
  Interventions: Drug: avanafil

INTERVENTIONS:
Drug: avanafil — 200 mg avanafil tablet QD

SUMMARY:
The objective of this study is to compare the pharmacokinetics of avanafil in subjects with mild and moderate renal impairment and to assess the safety and toleration of avanafil in subjects with mild and moderate renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Adult male subjects,
* 21-78 years of age, must be medically healthy with no clinically significant screening results (except for the subjects in Groups 2 and 3).
* Subjects with normal renal function (Group 1) must have an estimated CLcr of ≥80 mL/min.
* Subjects with renal impairment (Groups 2 and 3) must fulfill the additional following criteria: (a) Stable renal impairment; (b) Group 2 subjects with mild renal impairment must have a CLcr of ≥50 to <80 mL/min and (c) Group 3 subjects with moderate renal impairment must have a CLcr of ≥30 to <50 mL/min.

Exclusion Criteria:

* Major exclusion criteria include: history or clinical evidence of clinically relevant cardiovascular (including thromboembolic disorders), hepatic, renal (with the exception of renal insufficiency for subjects in Groups 2 and 3), hematological, endocrine, pulmonary, gastrointestinal, psychiatric or neurological impairment; any clinically significant laboratory abnormalities as judged by the Investigator; systolic blood pressure < 90 or >160 mmHg; diastolic blood pressure < 50 or > 95 mmHg; allergy to or previous adverse events with PDE5 inhibitors or its constituents; use of prescription or over-the-counter drugs that are known to interfere with metabolism by the cytochrome P450 3A4 enzyme within 30 days prior to Day 1; use of any investigational drug within 30 days prior to Day 1; use of any prescription or over-the-counter drugs or herbal remedies within 14 days prior to Day 1; history of alcohol or drug abuse within 18 months, history of smoking within 6 months; positive breathe alcohol test; positive cotinine test, positive urine drug screen (except in renally impaired subjects following approval by Sponsor). Additional exclusion criteria are listed in Section 4.2.

Ages: 21 Years to 78 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Single dose PK of avanafil | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Shiyin Yee, Study Director — VIVUS LLC